CLINICAL TRIAL: NCT04690036
Title: Reactivation of EBV for Patients With CAEBV and EBV Associated HLH After Transplantation
Brief Title: PD-1 Antibody for Reactive EBV After BMT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Department of Hematology, Beijing Friendship Hospital, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1,reactive EBV
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: PD-1; EBV Infection; Transplant
MeSH Terms: conditions — Epstein-Barr Virus Infections | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- one group (Experimental): All patients encountered EBV reactivation after allo-HCT could be enrolled in this study, there was only one group of treatment.
  Interventions: Drug: toripalimab injection

INTERVENTIONS:
Drug: toripalimab injection — when EBV-DNA is positive after allo-HCT, and EBV infected T/NK cell, one dose of toripalimab 3mg/kg would be used, the same dose would be repeated 4 weeks later.
  Other Names: EBV-DNA positive

SUMMARY:
PD-1 antibody for reactivation of EBV after transplantation in patients with CAEBV/EBV-HLH

DETAILED DESCRIPTION:
Transplantaion is recongnized as a cure for CAEBV and EBV associated HLH，however, many patients undergo the reactivation of EBV after transpaltion, patiens may at high risk for recurrence of the disease. PD-1 is a promising therapy to solve this problem.

The present study was a one-arm clinical study, the main subject is to evaluate the effect of PD-1 antibody on the clearance of EBV

ELIGIBILITY:
Inclusion Criteria:

1. Meet hemophagocytic lymphohistiocytosis (HLH)-04 diagnostic criteria; EBV-DNA in peripheral blood or EBER in tissue were positive, patients were diagnosed with EBV associated HLH (EBV-HLH). Chronic active EBV infection (CAEBV) was diagnosed by WHO criteria.
2. Undergo allo-HCT, have achieved full chimerism
3. Age >18 years old, gender is not limited.
4. After transplantation, EBV was reactivated and EBV-DNA was positive in blood
5. No secondary graft failure. (After grafted, ANC <0.5*10^9/l,PLT <10*10^9/l)
6. No uncontrollable infection
7. Withdraw immunosuppressor, no graft-versus-host disease was observed.
8. Before the start of the study, aminopherase (ALT/AST) and total bilirubin were normal. Serum creatinine ≤ 1.5 times the upper limit of Normal (ULN); No thyroid dysfunction. The left ventricular ejection fraction (LVEF) was normal.
9. Informed consent.

Exclusion Criteria:

1. Allergic to toripalimab
2. Serious immunoreaction: myocardial damage, hepatitis, pneumonia
3. Central nervous system symptoms
4. Serious mental illness;
5. Active bleeding of the internal organs
6. Pancreatitis history. Patients unable to comply during the trial and/or follow-up phase;
7. Participate in other clinical research at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
EBV-DNA turn negative | 4 weeks after PD-1 antibody was used
  after treatment, the EBV-DNA copies can not be detected in peripheral blood

SECONDARY OUTCOMES:
treatment-related adverse events as assessed by CTCAE v5.0 | 4 weeks after PD-1 antibody was used
  Adverse events including thyroid function，liver function damage, myelosuppression, infection, bleeding and so on

OTHER OUTCOMES:
Survival | 1 year
  From enrollment until death or the end of the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No